CLINICAL TRIAL: NCT06441539
Title: Bingo Drug-eluting Balloon Versus a Drug-eluting Stent for Coronary Bifurcation Lesions: a Prospective, Multi-center, Randomized, Non-inferiority Trial
Brief Title: Bingo Drug-eluting Balloon Versus a Drug-eluting Stent for Coronary Bifurcation Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yinyi(Liaoning) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNYY2024001
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary bifurcation; Percutaneous coronary intervention; Drug-coated balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug-eluting balloon (Experimental): Treat the main vessel and side branch of bifurcation lesion with drug-eluting balloon
  Interventions: Device: Bingo® Paclitaxel coated balloon
- drug-eluting stent (Active Comparator): Treat the main vessel of bifurcation lesion with drug-eluting stent, and treat the side branch with uncoated balloon or drug-eluting stent
  Interventions: Device: Xience® Alpine Everolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: Bingo® Paclitaxel coated balloon — Treat the main vessel and side branch of bifurcation lesion with drug-eluting balloon
  Arms: drug-eluting balloon
Device: Xience® Alpine Everolimus Eluting Coronary Stent System — Treat the main vessel of bifurcation lesion with drug-eluting stent, and treat the side branch with uncoated balloon or drug-eluting stent
  Arms: drug-eluting stent

SUMMARY:
Bingo drug-eluting balloon versus a drug-eluting stent for coronary bifurcation lesions: a prospective, multi-center, randomized, non-inferiority trial

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Age 18 to 80
2. Patients with chronic stable coronary artery disease, or unstable angina, or NSTEMI (Grace score<140), or STEMI more than one week
3. Subjects suitable for PCI
4. Subjects understand the trial purpose, volunteer to participate and sign informed consent form

Angiographic Inclusion Criteria (by visual):

1. One coronary de novo bifurcation lesion (including Medina classification: 1,1,1 / 1,0,1 / 0,1,1, which need to be treated for both main and side branches)
2. The reference vessel diameter of main branch is between 2.5 to 4.0 mm, length ≤ 30 mm. Before lesion preparation, lesion diameter stenosis shall be ≥70%, or ≥50% with evidence of myocardial ischemia
3. The reference vessel diameter of side branch is ≥2.0 mm, length <20 mm. Before lesion preparation, lesion diameter stenosis shall be ≥70%
4. No more than 3 lesions on the non-target vessel in the same operation, and shall be successfully treated before the target vessel
5. No more than 1 non-target lesion on the target vessel in the same operation, and shall be successfully prepared before the target lesion (successful preparation of non-target lesion is defined as residual stenosis ≤30% and TIMI flow 3). After randomization, the non-target lesion shall be treated according to the assigned group, for the experimental group, using the experimental DCB is recommended; for the control group, using DES is recommended; Independent lesion on the same coronary artery is defined as interval >5 mm
6. The target lesions of main and side branches must be successfully prepared (successful preparation is defined as: residual stenosis ≤30% , without NHLBI type C or above dissection, and TIMI flow 3)

Clinical Exclusion Criteria:

1. Severe heart failure (NYHA IV), cardiogenic shock or severe valvular heart disease
2. Left ventricular ejection fraction ≤35%
3. Severe renal insufficiency (eGFR <30 ml/min)
4. Severe liver insufficiency (glutamate transaminase (ALT) or glutamate transaminase (AST) >3 times the upper limit of normal)
5. Pregnant women or planned pregnancy
6. With a known allergy to heparin, contrast agent, paclitaxel and everolimus
7. Unable to receive antiplatelet agents and anticoagulants, bleeding tendency or coagulopathy
8. Life expectancy does not exceed 1 year
9. Participating in other drug or device clinical trials without reaching the primary endpoint
10. Subjects who had undergone coronary revascularization in the last 6 months
11. Subjects not eligible by the investigator for other reasons

Angiographic Exclusion Criteria (by visual):

1. In-stent restenosis lesion
2. Left main bifurcation lesion
3. Chronic total occlusive lesion
4. Target vessel is severely distorted, angulated or calcified, which is anticipated difficult to cross for balloon or stent
5. Target lesion remains significant residual thrombus after preparation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
in-segment late lumen loss in main branch | 9 months
  use quantitative coronary angiography by an independent core laboratory

SECONDARY OUTCOMES:
Procedure success rates | up to 7 days in-hospital
  include device success, lesion success and clinical success
Minimal lumen diameter | 9 months
  use quantitative coronary angiography by an independent core laboratory
Diameter stenosis | 9 months
  use quantitative coronary angiography by an independent core laboratory
Dissection and type | 9 months
  use quantitative coronary angiography by an independent core laboratory
in-segment late lumen loss in side branch | 9 months
  use quantitative coronary angiography by an independent core laboratory
Binary restenosis | 9 months
  use quantitative coronary angiography by an independent core laboratory
Target lesion failure | 1, 6, 9 and 12 months
  include cardiac death, target vessel myocardial infarction, clinically driven target lesion revascularization
Target lesion thrombosis | 1, 6, 9 and 12 months
  include acute, sub-acute, late and very late period
BARC bleeds | 1, 6, 9 and 12 months
  type 2, 3 or 5
Stroke | 1, 6, 9 and 12 months
  any stroke
Myocardial infarction | Peri-operation and 12 months
  include peri-operation and 12 months
Death | 1, 6, 9 and 12 months
  include cardiac and all-cause death
Major Adverse Cardiovascular Events | 1, 6, 9 and 12 months
  composite endpoint with death, myocardial infarction and target vessel revascularization